CLINICAL TRIAL: NCT05946473
Title: Development of a Novel Anti-caries Chewing Gum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Dennis Cvitkovitch, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 44196
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Dental Plaque; Dental Caries; Periodontal Disease
MeSH Terms: conditions — Dental Plaque; Dental Caries; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental gum formulation (Experimental): Participants will be asked to chew 2 pieces of chewing gum containing additives 2 times a day for a four-week period
  Interventions: Dietary Supplement: Gum base containing xylitol and essencial oils
- Placebo (Placebo Comparator): Participants will be asked to chew 2 pieces of pure gum base with no additives chewing gum 2 times a day for the same four-week period.
  Interventions: Dietary Supplement: Gum base with no additives

INTERVENTIONS:
Dietary Supplement: Gum base containing xylitol and essencial oils — Participants will be asked to chew 2 pieces of chewing gum containing additives for 10 minutes after eating in the morning, and after one meal in the evening, for a four-week period
  Arms: Experimental gum formulation
Dietary Supplement: Gum base with no additives — Participants will be asked to chew 2 pieces of pure gum base for 10 minutes after eating in the morning, and after one meal in the evening, for a four-week period
  Arms: Placebo

SUMMARY:
This research study is designed to evaluate the chewing gum's ability to modulate the oral microbiome in human participants, in addition to its safety.

DETAILED DESCRIPTION:
The goal of this project is to develop a pre-biotic chewing gum that is designed to promote a healthy oral microbiome. The gum will contain compounds that will: a) be unable to be converted to acids; b) target the cariogenic S. mutans population; c) promote the stability of a healthy environment by modulating plaque pH via base-generating compounds; d) promote tooth remineralization by increasing saliva flow and by addition of calcium phosphate.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, no relevant medical history
* No dental treatment in the previous 3 months
* Willing to participate and give written informed consent

Exclusion Criteria:

* Patients undergoing fixed or removable orthodontic treatment
* Patients using removable prosthesis
* History of head and neck radiation therapy
* History of adverse reaction or allergies to xylitol or other additives
* Antibiotics use in the last four weeks
* Patients with any systemic diseases
* Xerostomia (also medication-induced)
* Smokers
* Currently using any mouth rinse
* Pregnant or breastfeeding women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in target species of the oral microbiome | 28 days
  Total microbiome analyses will be performed at the beginning and end of the study (4 weeks) to assess total cultivable flora, levels of S. mutans, S. salivarius, and P. gingivalis in addition to using qRT-PCR from plaque and saliva samples